CLINICAL TRIAL: NCT05757817
Title: Evaluation of the Benefit of a New Surgical Procedure According to IDEAL Recommendations for ORL Cancer Patients: the External Pudendal Flap Used as a New Free Flap for Oral Cavity/Oropharyngeal Reconstruction to Limit Donor Site Sequelae
Acronym: LAMBEAU STEPA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 22VADS02
Record Dates: First submitted 2023-02-24; First posted 2023-03-07 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Head and Neck Cancer; Oral Cavity Cancer; Oropharynx Cancer
Keywords: Head and Neck Cancer; Oral Cavity Cancer; Oropharynx Cancer; STEPA flap; Oropharyngeal or oral cavity reconstruction; IDEAL Recommendations
MeSH Terms: conditions — Head and Neck Neoplasms; Mouth Neoplasms; Oropharyngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient with an ORL Cancer (Experimental)
  Interventions: Procedure: Oropharyngeal or oral cavity reconstruction

INTERVENTIONS:
Procedure: Oropharyngeal or oral cavity reconstruction — Oropharyngeal or oral cavity reconstruction will be performed using a free super thin external pudendal artery flap (STEPA flap).
  Post-operative follow-up and adjuvant treatment: Post-operative follow-up of patients will be performed according to the standards of the participating centers.

SUMMARY:
This is a phase 1b, multicenter, non-randomized prospective study involving an innovation phase (IDEAL-1) followed by a prospective development phase (IDEAL-2A) designed to evaluate the safety and feasibility of oral/oropharyngeal reconstruction with the external pudendal free flap in two groups of patients.

A maximum of 40 patients (20 patients per group) will be included in this IDEAL-1/2A phase study.

Stage IDEAL-1: Innovation phase. The main objective is to evaluate the feasibility in terms of limiting surgical complications of a STEPA flap reconstruction in two groups of patients (Cohort: Male, Female).

Stage IDEAL-2A: Prospective development phase. The main objective is to describe the complication profile of the surgical procedure in these two patient populations.

Each patient will be followed during 12 months after the end of complete treatment (surgery ± adjuvant treatment).

A complementary study (observational study) of 250 patients will also be conducted to evaluate the acceptability of the technique (reconstruction by external pudendal flap) by the patients and to describe the factors associated with this acceptability.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with a histologically proven diagnosis of head and neck squamous cell carcinoma (HNSCC) of the oral cavity or oropharynx.
2. Patient whose disease is classified UICC TNM stade (8th edition) : T0-4a N0/N2c M0 (no distant metastasis M0).
3. Patient whose oral cavity or oropharynx reconstruction requires a free fasciocutaneous flap according to an experienced oncology surgeon.
4. Patient OMS 0-1.
5. Age ≥ 18.
6. Patient with no contraindication to surgery.
7. Patient affiliated to a Social Health Insurance in France.
8. Patient able to participate and willing to give informed consent prior performance of any study-related procedures and to comply with the study protocol.

Exclusion Criteria:

1. Patient with history of prior cervical surgery and/or radiation to the head and neck.
2. History of pelvic surgery and/or radiation to the pelvic area.
3. Patients with a contraindication to any form of sedation.
4. Patient with irreversible coagulopathy.
5. Patient with a contraindication to a CT scan or an injection of iodinated contrast medium.
6. Patient with active autoimmune disorders requiring immunosuppressive therapy, defined as receiving steroids (dose > 10 mg of prednisone or equivalent) or other immunosuppressive therapy.
7. Pregnant or breastfeeding women.
8. Patient with another co-existing malignancy at the time of inclusion or any other significant medical, psychiatric, or surgical condition currently not controlled by treatment, which may interfere with the conduct of the study.
9. Patient with diabetes (type 1 or 2).
10. Patient with a BMI > 30kg/m².
11. Any psychological, family, geographic or sociological condition that does not allow for compliance with the medical follow-up and/or procedures provided for in the study protocol .
12. Patient who has forfeited his/her freedom by administrative or legal award or who is under legal protection (curatorship and guardianship, protection of justice).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
The occurrence of a limiting complication. Limiting complications are defined as total flap necrosis (flap failure) or donor site infection (Fournier Gangrene) within 4 weeks of the experimental procedure. | 4 weeks for each patient

SECONDARY OUTCOMES:
The postoperative complications will be evaluated according to the NCI-CTCAE version n°5 | 12 months for each patient
The pain will be assessed according to a Likert scale between 0 (no pain) and 10 (worst pain). | 12 months for each patient
The functional capacity of swallowing will be assessed via the Performance Status Scale for Head and Neck cancer patients - PSS-HN (Scales are: Normalcy of Diet, Public Eating, and Understandability of Speech). | 12 months for each patient
4. The aesthetic evaluation will be performed according to a Likert scale (Likert scale: not at all satisfied, somewhat not satisfied, neither dissatisfied nor satisfied, somewhat satisfied, very satisfied). | 12 months for each patient

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Chu Gui de Chauliac, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Chu Purpan, Toulouse
  - Institut Universitaire Du Cancer Toulouse - Oncopole (Iuct-O), Toulouse